CLINICAL TRIAL: NCT02106052
Title: The Effect of Aerobic Exercise on Cognition in Multiple Sclerosis (MS Exercise Study)
Brief Title: Study of Exercise on Impact of Cognitive Functioning in Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Charles Bombardier, Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46598
Record Dates: First submitted 2014-03-14; First posted 2014-04-07 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: cognitive function; cognitive impairment; cognitive intervention; cognitive improvement; information processing speed; exercise training program; aerobic exercise; stretching and toning; Multiple sclerosis; executive function
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Active Comparator)
  Interventions: Other: Aerobic exercise
- Stretching and toning exercise (Other)
  Interventions: Other: Stretching and toning exercise

INTERVENTIONS:
Other: Aerobic exercise — The aerobic exercise condition is a graduated program of supervised aerobic exercise up to one hour per day, three days per week, and lasting 6 months. The structured exercise portion of the sessions will initially last for 15-20 minutes at 40-50% heart rate reserve (HRR) and progressively increase up to 35-40 minutes in duration at 65-75% HRR during the last month of the program. The program will focus on large, dynamic movements of the lower extremities (e.g. leg cycling ergometry). There may be some individual variation in adaptations that dictate the exact characteristics of the program.
  Arms: Aerobic exercise
Other: Stretching and toning exercise — The stretching and toning condition is a supervised stretching program with Therabands up to one hour per day, three days per week, and lasting 6 months. The stretching exercises will be based on a manual published by the National Multiple Sclerosis Society (NMSS) that has been standardized, manualized for reproducibility, and the investigators will progressively include more exercises and sets with Therabands for resistance over the course of the 6-month period.
  Arms: Stretching and toning exercise

SUMMARY:
Cognitive impairment affects roughly 50% of people with multiple sclerosis (MS). There are currently no satisfactory medical treatments for cognitive impairments related to MS and alternative forms of treatment are needed. Exercise training can improve cognition in older adults and people with mild cognitive impairments, including those with early Alzheimer's disease. Therefore, the investigators plan to conduct the first definitive study that will test the theory that moderately intense aerobic exercise can improve cognition in people with MS-related impairment - specifically in information processing speed - more so than non-aerobic stretching and toning (both forms of exercise will be performed 3 days per week for 6 months).

Primary study hypothesis: The investigators hypothesize greater improvement in speed of information processing from pre- to post-treatment in the aerobic exercise group compared to the stretching and toning group (attention control).

Secondary study hypothesis: The investigators hypothesize greater improvement in other cognitive domains and patient reported outcomes from pre- to post-testing in the aerobic exercise group compared to the stretching and toning group (attention control).

The investigators plan to recruit 125 adults with MS who can walk without assistance and without rest for at least 100 meters and have mild weaknesses in information processing speed. The investigators will randomly assign 50% of participants to an aerobic exercise program and 50% to a non-aerobic exercise program (stretching and toning). In order to determine whether the intervention is successful, the investigators will compare cognitive functioning in both exercise groups before the exercise-training program, at the end of the 6-month training program and three months after the end of the training program. If our study findings support our hypotheses, this would be a relatively no-barriers treatment option to further explore for other people with MS including people with greater and lesser baseline disability.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language.
* At least 9th grade education.
* Physician confirmed, clinically definite MS diagnosis as defined by the revised McDonald criteria.
* All MS subtypes will be included.
* MS diagnosis at least 6 months prior.
* Impaired speed of information processing and working memory based on either the PASAT-3" or the SDMT (i.e. z <-1.5 controlling for age, education and sex).
* Physician clearance to engage in aerobic exercise training.
* Able to walk at least 100 meters without assistance (Expanded Disability Severity Scale score equivalent 0-5.5).
* Currently exercising less than public health recommendations (engaging in less than 30 minutes of structured physical activity less than 3 times per week during the past 6 months).
* Willingness not to undertake additional structured exercise or leisure time physical activity during the 6-month trial.
* Willing and able to participate in either exercise training program 3 days per week for 6 months at a YMCA in the Greater Seattle Area.

Exclusion Criteria:

* Near visual acuity with correction 20/70 or worse.
* Contra-indications for exercise training based on American Heart Association (AHA)/ACSM screening criteria using PAR-Q.
* Using any medication known to have adverse effects on motor or cognitive function, including monoamine oxidase inhibitors, sympathomimetics, antipsychotic agents, modafinil, oxybutynin, tricyclic antidepressants, cholinesterase inhibitors and anticonvulsants other than gabapentin and pregabalin. The following are permitted if the patient has been on a stable dose for at least 6 weeks: short acting benzodiazepines (qhs administration only), anti-spasmodics, selective serotonin reuptake inhibitors and serotonin-norepinephrine reuptake inhibitors.
* Received steroids in last 30 days.
* Relapse in the last 90 days.
* Undergone neuropsychological testing within the past 6-months.
* Neurological/psychological disease other than MS that may impact cognitive status, e.g. Alzheimer's disease, Parkinson's, stroke, TIA, Vascular Dementia, Huntington's, traumatic brain injury or chronic CNS infection.
* Dementia based on a definition validated in people with MS using the MACFIMS (> 2 SD below the mean on at least one memory test and > 2 SD below the mean on at least one neuropsychological test in another domain).
* Prior history of diagnosis or treatment for serious mental illness (obsessive-compulsive disorder, schizophrenia, other psychotic disorders, bipolar disorder).
* Diagnosis of major depressive disorder prior to the diagnosis of MS.
* History of significant developmental or learning disorder that may affect participation and confound interpretation of study results.
* Current major depressive disorder.
* Current alcohol or other drug abuse as measured by the WHO Alcohol, Smoking and Substance Involvement Screening Test (WHO ASSIST V3.0).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Composite score of the Paced Auditory Serial Addition Test-3 (PASAT-3") and the oral version of the Symbol-Digit Modalities Test (SDMT) | Baseline and six months after baseline.
  The PASAT-3" is an auditory processing speed measure in which patients are exposed to single digit numbers voiced every three seconds. After each number presentation, the patient's task is to respond with the sum of the last two digits presented. There are 60 stimuli. The main score is the number of correct responses. The SDMT will be used to measure visual processing speed. This test presents a stimulus key of numbers paired with abstract symbols at the top of a page. Patients scan the page below the key that has rows of symbols without the paired numbers. The task is to generate the associated numbers orally as fast as possible.

SECONDARY OUTCOMES:
Delis Kaplan Executive Function System Sorting Test (DKEFS) | The DKEFS will be administered at six months after baseline.
  The DKEFS will be used to assess higher executive function. Six cards are presented which can be sorted in at least eight different ways (e.g., card color, card shape, semantic association). Patients are allowed four minutes with each deck to sort the cards in as many ways possible. The dependent variables are the total number of correct sorts and the total verbal description score among the two decks.
California Verbal Learning Test, second edition (CVLT2) | The CVLT2 will be administered at six months after baseline.
  The CVLT2 will be used to evaluate multi-trial learning and long-term recall for verbal information. The test presents a list of 16 words over 5 learning trials using a selective reminding procedure. Patients are asked to recall as many words as they can after each trial followed by a delay interval, after which they are again asked to recall as many words from the list as possible. The investigators will use the total number of words recalled during the initial learning trials and the number of words recalled after the delay interval as outcomes for this study.
Brief Visuospatial Memory Test Revised (BVMTR) | The BVMTR will be administered at six months after baseline.
  The BVMTR will be used to assess visuospatial memory. The test presents a matrix of six visual designs over three learning trials, each time for 10 seconds. After each trial the patient is asked to reproduce the figures in their correct location. After a 20-25 minute delay, patients are again asked to redraw the designs. The investigators will use the total score over the three learning trials and the total number recalled after the 20-25 minute delay as outcomes.
The Controlled Oral Word Association Test (COWAT) | The COWAT will be administered at six months after baseline.
  The COWAT will be used to assess verbal fluency. The test requires patients to generate words orally that begin with a given letter of the alphabet. The outcome is the total number of correct words over the three trials.

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Bombardier, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Bombardier CH, Motl RW, Benedict RHB, Temkin N, Qian P, Alexander K, Evans A, Thomas A, Toms K, Carey CM, Kraft GH. Exercise training and cognition in multiple sclerosis: The GET Smart trial protocol. Contemp Clin Trials. 2021 May;104:106331. doi: 10.1016/j.cct.2021.106331. Epub 2021 Feb 27. PMID 33652128